CLINICAL TRIAL: NCT06902519
Title: A Phase 1b, Randomized, Blinded, Placebo-Controlled, Multicenter Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of GS-0151 in Adult Participants With Rheumatoid Arthritis
Brief Title: Study of GS-0151 in Participants With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-667-6882; 2024-516520-34 (Other: European Medicines Agency)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: In Part A, Cohorts 1 and 2 will be sequential, with participants receiving treatment in parallel and randomized in 6:2 ratio to either GS-0151 or placebo. In Part B, Cohort 3 will also randomized in 2:1 ratio to receive GS-0151 or placebo in parallel.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Cohort 1 (GS-0151 Dose A) (Experimental): Participants with RA will be randomized to receive Dose A of GS-0151 up to 12 weeks.
  Interventions: Drug: GS-0151
- Part A: Cohort 1 (Placebo) (Placebo Comparator): Participants with RA will be randomized to receive placebo up to 12 weeks.
  Interventions: Drug: Placebo
- Part A: Cohort 2 (GS-0151 Dose B) (Experimental): Participants with RA will be randomized to receive Dose B of GS-0151 up to 12 weeks.
  Interventions: Drug: GS-0151
- Part A: Cohort 2 (Placebo) (Placebo Comparator): Participants with RA will be randomized to receive placebo up to 12 weeks.
  Interventions: Drug: Placebo
- Part B: Cohort 3 (GS-0151 Dose C) (Experimental): Participants with moderately to severely active RA will be randomized to receive Dose C of GS-0151.
  Interventions: Drug: GS-0151
- Part B: Cohort 3 (Placebo) (Placebo Comparator): Participants with moderately to severely active RA will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-0151 — Administered for 12 weeks
  Arms: Part A: Cohort 1 (GS-0151 Dose A); Part A: Cohort 2 (GS-0151 Dose B); Part B: Cohort 3 (GS-0151 Dose C)
Drug: Placebo — Administered for 12 weeks
  Arms: Part A: Cohort 1 (Placebo); Part A: Cohort 2 (Placebo); Part B: Cohort 3 (Placebo)

SUMMARY:
The goal of this clinical study is to learn more about the study drug GS-0151. The study is done to find how safe, well-tolerated the drug is. This will also assess how the drug is absorbed, modified, distributed and cleared from the body (the pharmacokinetics (PK) of the drug), when given multiple times to participants with rheumatoid arthritis (RA).

The primary objectives of this study is to assess the safety and tolerability of multiple ascending doses of GS-0151 in participants with RA and to characterize the PK of GS-0151 following multiple doses of GS-0151 in participants with RA.

ELIGIBILITY:
Key Inclusion Criteria:

Medical History/Physical Characteristics; All Cohorts:

* Individuals must not be on a biologic disease-modifying antirheumatic drug (b/tsDMARD) on Day 1 and must have discontinued all b/tsDMARDs (including biosimilars and generics) at least 4 weeks prior to Day 1 with the exception of B cell-depleting agents (eg, rituximab), which must be discontinued for at least 6 months prior to Day 1.
* Ongoing treatment with at least 1 but no more than 2 protocol-permitted conventional synthetic disease-modifying antirheumatic drug (csDMARDs) for at least 12 weeks, at a stable dose for at least 6 weeks prior to Day 1 and remain stable throughout the treatment period:

  1. Use of oral, intramuscular (IM), or subcutaneous(ly) (SC) methotrexate 7.5 to 25 mg/week. Individuals on methotrexate must be receiving folic or folinic acid supplementation at a stable dose.
  2. Oral hydroxychloroquine ≤ 400 mg/day or chloroquine ≤ 250 mg/day.
  3. Oral sulfasalazine 1 to 3 g/day.
  4. Oral leflunomide 10 to 20 mg/day.
* Use of oral corticosteroids of no more than 10 mg prednisone or equivalent per day is allowed if the dose is stable for at least 14 days prior to Day 1. Inhaled corticosteroids for stable medical conditions are allowed but must have been at a stable dose for at least

  1 week prior to the first dose of study drug. Occasional topical corticosteroids are permitted.
* Where nonsteroidal anti-inflammatory drug (NSAIDs) or acetaminophen are used, the dose must be stable for at least 1 week prior to Day 1
* Individuals must have discontinued all high-potency opiates at least 1 week prior to Day 1.

Cohort 3 Only:

* Individuals must meet all of the following cohort-specific inclusion criteria, in addition to meeting the inclusion criteria for all individuals , to be eligible for participation in Part B:

Moderately to severely active RA defined by the following:

Screening and Day 1:

1. 6 or more tender joints on the tender joint count based on 68 joints (TJC68), AND.
2. 6 or more swollen joints on the swollen joint count based on 66 joints (SJC66). The distal interphalangeal joints should be evaluated but not included in the total count to determine eligibility.

   Screening Only
3. Have a hsCRP ≥ ULN

   * Inadequate response or intolerance to at least 1 but no more than 3 b/tsDMARDs with no more than 2 mechanisms of action. A lack of response is defined as documented continued or recurrent disease activity after at least 12 weeks of treatment of RA. Intolerance is defined as any documented adverse effect associated with a b/tsDMARD used according to its respective label.

Laboratory Assessments:

Cohort 3 Only:

* Anti-cyclic citrullinated peptide antibody (Anti-CCP) positive and/or rheumatoid factor (RF) positive

Key Exclusion Criteria:

Medical Conditions; All Cohorts:

* Have a diagnosis of any generalized musculoskeletal disorder that would interfere with study procedures or assessments per the discretion of the investigator.
* History of opportunistic infection or immunodeficiency syndrome that would put the individual at risk, as per investigator's judgment.
* Active infection that is clinically significant, per investigator's judgment, or any infection requiring hospitalization or treatment with intravenous anti-infectives within 60 days of screening; or any infection requiring oral anti-infective therapy within 30 days of screening.
* History of or current moderate to severe congestive heart failure (New York Heart Association class III or IV), or within the last 6 months prior to screening.
* History of lymphoproliferative disease or possible current lymphoproliferative disease.
* History of organ or bone marrow transplant.
* Have a history of major surgery (requiring regional block or general anesthesia) within the last 12 weeks prior to screening or planned major surgery during the study.
* History of an infected joint prosthesis or other implanted device with the prosthesis or device still in situ.
* Clinically significant ECG abnormalities at screening, including electrocardiographic interval between the beginning of the Q wave and termination of the T wave, representing the time for both ventricular depolarization and repolarization to occur (QT) interval corrected for heart rate using the Fridericia formula (QTcF) > 450 msec, or hypokalemia if recurrent or persistent < 3.0 mmol/L, or family history of long QT syndrome

Prior/Concurrent Therapy or Clinical Study Experience:

* Administration of a live attenuated vaccine 4 weeks prior to Day 1 or planned throughout the study.
* Participation in any investigational drug/device clinical study within 4 weeks or 5 half-lives prior to screening, whichever is longer. Exposure to investigational biologics should be discussed with the sponsor.

Diagnostic Assessments; All Cohorts:

* Any positive tuberculosis (TB) test using interferon-gamma release assay (IGRA) performed by central laboratory at screening. Tests with inconclusive results may be repeated one time. If an inconclusive test is repeated and is returned with inconclusive results a second time, the individual will be excluded from the study. Individuals with a history of latent or active TB who have been treated with a full course of treatment, as per local guidelines, are eligible without the need for an IGRA at screening. Appropriate documentation of prior treatment is required.
* Evidence of active hepatitis C virus (HCV) infection. Individuals with positive HCV Ab at screening require reflex testing for HCV ribonucleic acid (RNA). Individuals with positive HCV Ab but negative HCV RNA viral load are eligible per investigator judgment and require HCV viral load monitoring on Day 85 and Day 169.
* The results of the following laboratory tests performed at the central laboratory at screening meet any of the criteria below (out-of-range laboratory values may be rechecked 1 time, per investigator's judgment, before individual is considered a screen failure):

  1. Hemoglobin < 10.0 g/dL (SI: < 100 g/L)
  2. White blood cells < 3.0 x 10^3 cells/mm^3 (SI: < 3.0 x 10^9 cells/L)
  3. Neutrophils < 1.5 x 10^3 cells/mm^3 (SI: < 1.5 x 10^9 cells/L)
  4. Lymphocytes < 1.0 x 10^3 cells/mm^3 (SI: < 1.0 x 10^9 cells/L)
  5. Platelets < 100 x 10^3 cells/mm^3 (SI: < 100 x 10^9 cells/L)
  6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 x upper limit of normal (ULN)
  7. Total bilirubin level ≥ 2 x ULN unless the individual has been diagnosed with Gilbert's disease and this is clearly documented
  8. Creatinine clearance < 50 mL/min (SI: < 0.83 mL/s) based on the Cockcroft-Gault formula

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Cohort 1, 2 and 3: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) | First dose up to 19 Weeks post end of treatment at Week 12
Cohort 1, 2 and 3: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities | First dose up to 19 Weeks post end of treatment at Week 12
Cohorts 1, 2 and 3: Percentage of Participants Experiencing Serous Adverse Events (SAEs) and Adverse Events (AEs) Leading to Study Discontinuation | First dose up to 19 Weeks post end of treatment at Week 12
Cohort 1, 2 and 3: Serum AUCtau Following the Last Dose of GS-0151 | Up to Week 12
  AUCtau is defined as the area under the serum concentration versus time curve over the dosing interval.
Cohorts 1, 2 and 3: Serum Cmax, Following the Last Dose of GS-0151 | Up to Week 12
  Cmax is defined as the maximum observed plasma drug concentration.
Cohorts 1, 2 and 3: Serum Tmax Following the Last Dose of GS-0151 | Up to Week 12
  Tmax is defined as the time (observed time point) of Cmax.

SECONDARY OUTCOMES:
Cohorts 1, 2, and 3: Percentage of Participants with Antidrug Antibodies (ADAs) During the Study | Up to Week 12
Cohort 3: Change From Baseline in Disease Activity Score for 28 Joint Count Using C-Reactive Protein (DAS28-CRP) at Week 12 in Participants With Moderately to Severely Active RA | Baseline, Week 12
  The DAS28-CRP Score comprises tender joint count and swollen joint count based on a 28 joint assessment; patient's global assessment of disease activity and CRP. The DAS28-CRP Score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity), and hsCRP (CRP=hsCRP) for a total possible score of 1 to 9.4. Higher values indicate higher disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (32):
- United States (15):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of California, San Diego, La Jolla, California
  - Stanford University School of Medicine, Palo Alto, California
  - Medvin Clinical Research, Tujunga, California
  - Medvin Clinical Research, Whittier, California
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Great Lakes Clinical Trials dba Flourish Research Chicago, Chicago, Illinois
  - DM Clinical Research, Melrose Park, Illinois
  - Accurate Clinical Research, Inc, Lake Charles, Louisiana
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Accurate Clinical Research, Inc, Houston, Texas
  - Clinical Trials of Texas LLC, dba Flourish Research, San Antonio, Texas
  - Tidewater Clinical Research, LLC/ Virginia Rheumatology Clinic, Virginia Beach, Virginia
- ARENSIA Exploratory Medicine, LLC, Tbilisi, Georgia
- Germany (4):
  - Universitatsklinikum Koln, Cologne
  - Krakenhaus Porz am Rhein, Cologne
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Klinikum der Universitat Munchen, München
- Republican Clinical Hospital "Timofei Mosneaga," Arensia EM, Chisinau, Moldova
- Poland (6):
  - Clinicmed Daniluk, Bialystok
  - FutureMeds Gydinia, Gdynia
  - FutureMeds Lodz, Lodz
  - MICS Centrum Medyczne Torun, Torun
  - FutureMeds Targowek, Warszawa Targówek
  - FutureMeds Wroclaw, Wroclaw
- Spain (5):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitari Parc Tauli, Sabadell
  - Hospital Quironsalud Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06902519